CLINICAL TRIAL: NCT02280239
Title: Safety and Antipyretic Efficacy of Acetaminophen in the Febrile Intensive Care Unit Patient.
Brief Title: Safety and Efficacy of Acetaminophen in the Intensive Care Unit.
Acronym: SEA-ICU
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Only enrolled 10 participants over 9 months which is less then anticipated (75).
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health Research Institute (Other)
Responsible Party: Principal Investigator, Vininder K. Bains, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H13-01160
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Results first posted 2022-11-04 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Critical Illness; Fever
Keywords: Fever; Acetaminophen; Body Temperature Regulation; Critical Illness; Hypotension
MeSH Terms: conditions — Critical Illness; Fever; Hypotension | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): This group consists of stable but febrile ICU patients (temp >38.3°C). Participants in this group will receive a one-time dose of placebo via the enteral route (via the gut), after which vital signs (including continuous measures of core temperature, heart rate, and blood pressure) will be monitored for 4 hours.
  Interventions: Drug: Placebo
- Acetaminophen Group (Experimental): This group consists of stable but febrile ICU patients (temp >38.3°C). Participants in this group will receive a one-time does of acetaminophen 650mg via the enteral route (via the gut), after which vital signs (including continuous measures of core temperature, heart rate, and blood pressure) will be monitored for 4 hours.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — one-time dose of acetaminophen 650mg given via the enteral route (via the gut)
  Other Names: Tylenol
  Arms: Acetaminophen Group
Drug: Placebo — one-time dose of placebo (identical capsule) given via the enteral route (via the gut)
  Other Names: Pharmacy compounded look alike capsule to the study drug
  Arms: Control Group

SUMMARY:
The intensive care unit (ICU) team needs to know what effects acetaminophen has in critically ill patients. Acetaminophen is better known as Tylenol. It is the drug given to reduce fever. Most research that has looked at how safe and effective this drug is, has been done with healthy people. Those studies tell us it is safe and works well to bring down fever.

This may not be true for the ICU patient. Some research found acetaminophen was not as good at reducing fever as expected in the ICU. Fever helps to fight infection so it may help patients get better, but it is also stressful. When you have fever, you to need more oxygen, and your heart beats faster. If you have a fever after brain injury, you are less likely to make a full recovery. In patients with brain injury, a weak heart or trouble breathing we should treat fever. If we can predict how well acetaminophen will reduce fever, we can decide if this drug is enough, or other treatments are also needed.

If you do not have problems with your brain, heart, or lungs, it is safe to not treat fever. When you give this drug to treat fever, the body cools itself by sweating, and bringing hot blood to the skin's surface. These changes do not affect healthy people. Research suggests ICU patients may be at risk for sudden drop in blood pressure.

Our study will answer 2 questions: 1) When acetaminophen is given to treat fever in ICU patients, are they more likely to have a drop in blood pressure? 2) How much will acetaminophen reduce fever in ICU patients? We will study ICU patients with a fever who can safely get, or not get this drug. This information will help us decide when and how to treat fever in the ICU.

DETAILED DESCRIPTION:
In the ICU, fever is commonly treated with 650 mg acetaminophen every 4 hours with the hopes of reducing fever burden, thereby also reducing metabolic demand. Acetaminophen is thought to be a safe and effective antipyretic. This assumption has not been tested in the critically ill despite its widespread use. Observational studies report critically ill patients experience hypotension, sometimes severe enough to require treatment; other studies indicate acetaminophen may not be as effective at reducing fever burden in the critically ill.

OBJECTIVES:

* To see if 650mg acetaminophen, given to febrile critically ill patients affects blood pressure; by comparing the incidence of hypotension severe enough to require treatment in the way of a fluid bolus (500cc or greater) or increase in vasoactive drugs (increase in norepinephrine by 5mcg or greater); by assessing for changes in mean arterial pressure and systolic blood pressure.
* To quantify the degree of fever suppression achieved by 650mg acetaminophen in the febrile critically ill population.

RESEARCH PROPOSAL:

Patients admitted into Vancouver Hospital's ICU are eligible for this study if they have a new fever and meet the inclusion/exclusion criteria. Study participants will be randomly assigned into one of 2 study arms, the control group and the 650mg group. Study participants in the control group will receive 2 capsules of placebo and the 650mg group will receive 2 capsules of 325mg acetaminophen. Data (continuous measures of temperature, heart rate and blood pressure) will be collected from the time of the study drug administration until 6 hours post. All patients, health care workers, and researchers will be blinded to which arm the patient is enrolled in until the end of the study. The incidence of fluid bolus administration, increases in vasoactive drug use, will be recorded and compared. We will also compare blood pressure data, and fever burden between the 2 groups.

INCLUSION/EXCLUSION CRITERIA To be included the subject must be admitted to the ICU; have an arterial line as standard of care; have at least 2 hours of a temperature greater than 38.3°C; within 24 hours of fever onset or ICU admission; be hemodynamically stable, and not received any drugs with known antipyretic effects at least 6 hours prior to initiating the study. Patients are excluded if they have an acute brain injury, liver dysfunction, cardiac dysfunction, requiring greater than 50% fraction of inspired oxygen (FiO); mechanical ventilation is permitted, any extracorporeal blood treatments (dialysis, plasmapheresis, etc.), injury to more than 20% of the skin (i.e. burn patient), or the responsible physician is opposed to enrolment.

ELIGIBILITY:
Generally to be considered for this study one must be critically ill, febrile, and can safely either receive acetaminophen or have acetaminophen withheld. Also one must not have conditions that would alter normal drug absorption or normal thermoregulation. Specifically the eligibility criteria are:

INCLUSION CRITERIA:

* Adult patients (> 18 years) admitted to Intensive Care Unit at Vancouver Hospital with a core temperature > 38.3 °C for 2 or more consecutive hours, but not longer than 48 hours*
* Continuous arterial pressure monitor in place at the time of intervention and data collection
* Patients may only participate in the study once
* To remain in the ICU for the entire study period (2 hours prior to drug administration to 4 hours post drug administration)

EXCLUSION CRITERIA:

* Significant liver dysfunction
* Acute neurological injury
* Seizure disorder
* Cardiomyopathy, elevated cardiac enzymes indicative of an acute cardiac injury, electrocardiogram (ECG) changes indicative of cardiac ischemia (i.e., ST segment elevation/depression)
* Hemodynamic instability (requiring fluid boluses, or change/initiation of vasopressors. Patients receiving steady doses of vasopressor support may be included)
* Severe hypoxemia, (fraction of inspired oxygen (FiO2) requirements of more than 60% to maintain hemoglobin oxygen saturation (SaO2) > 90% or partial pressure of oxygen in the blood (PaO2) > 70)
* Temperature > 40.0 °C
* Receiving external cooling
* Haemodialysis, plasma exchange, or any treatment where the blood is taken out of the body and processed
* Acute thermal injury to skin (i.e., burn)
* Gut malabsorption (i.e., receiving < 40% required calories enterally)
* Receiving medications that have known antipyretic effects (acetaminophen, ibuprofen, steroids, etc.)
* Physician opposed to enrolment in the study

NOTE: in response to very low enrollment 2 exclusion criteria were changed on Nov 5, 2015. These were:

1. patients no longer needed to recieve 40% of required calories enterally, instead patients who were not receiving any caloric intake via the gut could be enrolled as long as they were still permitted to receive oral medications.
2. patients no longer had to have acetaminophen discontinued upon enrollment. They could not be receiving it regularly but could still receive acetaminophen on an as needed (PRN) basis as long as it could be safely withheld for up to 12 hours if they developed a fever.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Henderson, PhD, Study Chair — University of British Columbia; Vininder K Bains, BSN, Principal Investigator — Vancouver Coastal Health; Martha Mackay, PhD, Study Chair — University of British Columbia; Leanne Currie, PhD, Study Chair — University of British Columbia
Locations (1):
- Vancouver Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Under review with the research team.

REFERENCES:
- [Background] Russell JA, Walley KR, Singer J, Gordon AC, Hebert PC, Cooper DJ, Holmes CL, Mehta S, Granton JT, Storms MM, Cook DJ, Presneill JJ, Ayers D; VASST Investigators. Vasopressin versus norepinephrine infusion in patients with septic shock. N Engl J Med. 2008 Feb 28;358(9):877-87. doi: 10.1056/NEJMoa067373. PMID 18305265
- [Background] Finfer S, Bellomo R, Boyce N, French J, Myburgh J, Norton R; SAFE Study Investigators. A comparison of albumin and saline for fluid resuscitation in the intensive care unit. N Engl J Med. 2004 May 27;350(22):2247-56. doi: 10.1056/NEJMoa040232. PMID 15163774
- [Background] Vincent JL, Weil MH. Fluid challenge revisited. Crit Care Med. 2006 May;34(5):1333-7. doi: 10.1097/01.CCM.0000214677.76535.A5. PMID 16557164
- [Background] Boyle M, Nicholson L, O'Brien M, Flynn GM, Collins DW, Walsh WR, Bihari D. Paracetamol induced skin blood flow and blood pressure changes in febrile intensive care patients: An observational study. Aust Crit Care. 2010 Nov;23(4):208-14. doi: 10.1016/j.aucc.2010.06.004. Epub 2010 Jul 22. PMID 20655241
- [Background] Boyle M, Hundy S, Torda TA. Paracetamol administration is associated with hypotension in the critically ill. Aust Crit Care. 1997 Dec;10(4):120-2. doi: 10.1016/s1036-7314(97)70414-4. PMID 9708071
- [Background] Krajcova A, Matousek V, Duska F. Mechanism of paracetamol-induced hypotension in critically ill patients: a prospective observational cross-over study. Aust Crit Care. 2013 Aug;26(3):136-41. doi: 10.1016/j.aucc.2012.02.002. Epub 2012 Mar 14. PMID 22424816
- [Background] Allegaert K, Naulaers G. Haemodynamics of intravenous paracetamol in neonates. Eur J Clin Pharmacol. 2010 Sep;66(9):855-8. doi: 10.1007/s00228-010-0860-z. Epub 2010 Jul 4. PMID 20607221
- [Background] de Maat MM, Tijssen TA, Bruggemann RJ, Ponssen HH. Paracetamol for intravenous use in medium--and intensive care patients: pharmacokinetics and tolerance. Eur J Clin Pharmacol. 2010 Jul;66(7):713-9. doi: 10.1007/s00228-010-0806-5. Epub 2010 Mar 19. PMID 20300741
- [Background] Danguy des Deserts M, Nguyen BV, Giacardi C, Commandeur D, Paleiron N. [Acetaminophen-induced hypotension after intravenous and oral administration]. Ann Fr Anesth Reanim. 2010 Apr;29(4):313-4. doi: 10.1016/j.annfar.2010.02.006. Epub 2010 Mar 12. No abstract available. French. PMID 20227233
- [Background] Mrozek S, Constantin JM, Futier E, Zenut M, Ghardes G, Cayot-Constantin S, Bonnard M, Ait-Bensaid N, Eschalier A, Bazin JE. [Acetaminophene-induced hypotension in intensive care unit: a prospective study]. Ann Fr Anesth Reanim. 2009 May;28(5):448-53. doi: 10.1016/j.annfar.2009.01.018. Epub 2009 Mar 21. French. PMID 19304444
- [Background] Hersch M, Raveh D, Izbicki G. Effect of intravenous propacetamol on blood pressure in febrile critically ill patients. Pharmacotherapy. 2008 Oct;28(10):1205-10. doi: 10.1592/phco.28.10.1205. PMID 18823215
- [Background] Cruz P, Garutti I, Diaz S, Fernandez-Quero L. [Metamizol versus propacetamol: comparative study of the hemodynamic and antipyretic effects in critically ill patients]. Rev Esp Anestesiol Reanim. 2002 Oct;49(8):391-6. Spanish. PMID 12455318
- [Background] Mackenzie I, Forrest K, Thompson F, Marsh R. Effects of acetaminophen administration to patients in intensive care. Intensive Care Med. 2000 Sep;26(9):1408. doi: 10.1007/s001340000614. No abstract available. PMID 11089781
- [Background] Bendjelid K, Soubirou JL, Bohe J. [Systemic arterial hypotension induced by paracetamol administration: nurse's anecdotes or facts from the intensive care unit?]. Ann Fr Anesth Reanim. 2000 Jun;19(6):499. doi: 10.1016/s0750-7658(00)00230-6. No abstract available. French. PMID 10941454
- [Background] Gozzoli V, Treggiari MM, Kleger GR, Roux-Lombard P, Fathi M, Pichard C, Romand JA. Randomized trial of the effect of antipyresis by metamizol, propacetamol or external cooling on metabolism, hemodynamics and inflammatory response. Intensive Care Med. 2004 Mar;30(3):401-7. doi: 10.1007/s00134-003-2087-2. Epub 2004 Jan 13. PMID 14722642
- [Background] Greenberg RS, Chen H, Hasday JD. Acetaminophen has limited antipyretic activity in critically ill patients. J Crit Care. 2010 Jun;25(2):363.e1-7. doi: 10.1016/j.jcrc.2009.07.005. Epub 2009 Sep 24. PMID 19781895

RESULTS

PARTICIPANT FLOW:
Recruitment Details: SCREENING: Of the 950 patients who were admitted between May 28, 2015 and Jan. 20, 2016, 790 were screened, at least once. A few were screened a second time if their status had changed.
  ELIGIBILITY: 100 patients were eligible.
  RECRUITMENT: 27/100 were successfully contacted to be invited to this study. 10 consented to participate.
Pre-assignment Details: Of the 10 participants who were successfully recruited to the study, only 6 developed a fever while in the ICU and could be randomized into either the control or acetaminophen group
Groups:
- Control Group: TOTAL: 1 Stable, febrile (temp >38.3°C) ICU patient/participant.
  Placebo: one-time dose of placebo (identical capsule) given via the enteral route (via the gut) after which vital signs (including continuous measures of core temperature, heart rate, and blood pressure) will be monitored for 4 hours.
- Acetaminophen Group: TOTAL: 5 stable febrile (temp >38.3°C) ICU patients/participants.
  Acetaminophen: one-time dose of acetaminophen 650mg given via the enteral route (via the gut) after which vital signs (including continuous measures of core temperature, heart rate, and blood pressure) will be monitored for 4 hours.
Period: Overall Study
Arm/Group | Control Group | Acetaminophen Group
Started | 1 | 5
Completed | 1 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Acetaminophen Group | Total
Number analyzed (Participants) | 1 | 5 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 5 | 5
  >=65 years | 1 | 0 | 1
Age, Continuous [Median (Full Range); unit: years] | 76 [76 to 76] | 35 [29 to 59] | 43.5 [29 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Clinically Significant Hypotension
Description: Clinically significant hypotension is defined as an acute drop in mean arterial pressure requiring treatment. Treatment is defined as either a 500 cc (or greater) fluid bolus and/or an increase in inotrope support of greater than 5 mcg/min over baseline.
Time Frame: 4 hours post acetaminophen administration
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Acetaminophen Group
Number analyzed (Participants) | 1 | 5
Participants | 0 | 0

2. Secondary Outcome: Blood Pressure
Description: systolic blood pressure (SBP), diastolic blood pressure (DBP) and mean arterial pressures (MAP) will be monitored for 4 hours post intervention
Time Frame: 4 hours post intervention
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Control Group | Acetaminophen Group
Number analyzed (Participants) | 1 | 5
mmHg
  SBP: Pre-Intervention (2 hours) | 141.6 [102 to 159] | 122.6 [80 to 170]
  SBP: Post-Intervention (4 hours) | 141.5 [127 to 157] | 119.5 [86 to 158]
  DBP: Pre-Intervention (2 hours) | 57.4 [46 to 63] | 66.2 [45 to 91]
  DBP: Post-Intervention (4 hours) | 51.0 [47 to 55] | 65.4 [45 to 83]
  MAP: Pre-Intervention (2 hours) | 80.8 [61 to 90] | 84.1 [56 to 114]
  MAP: Post-Intervention (4 hours) | 75.5 [68 to 83] | 82.4 [61 to 107]

3. Secondary Outcome: Equivalent-dose of Vasoactive Medication Post Intervention
Description: Total dose of all vasoactive medications will be converted to total Equidose value (with the formula 10 mcg/min norepinephrine ≈ 5 mcg/kg/min dopamine ≈ 10 mcg/min epinephrine ≈ 1 mcg/min phenylephrine ≈ 0.02 u/min vasopressin as per Russell et al. (2008)) before comparing the treatment and control groups
  Only 2 of the 6 participants were on low-dose vasoactive medications, (i.e., one was on norepinephrine and the other was on milrinone) therefore the pre-planned conversion calculation was not done.
Time Frame: 4 hours post intervention
Population: no analysis was done because the participant in the control group received norepinephrine and only 1 participant in the acetaminophen received milrione
Measure: Number; unit: mcg
Groups:
- Control Group: TOTAL: 1 Stable, febrile (temp >38.3°C) ICU patient/participant.
  Placebo: one-time dose of placebo (identical capsule) given via the enteral route (via the gut) after which vital signs (including continuous measures of core temperature, heart rate, and blood pressure) will be monitored for 4 hours.
  This participant was on a low dose norepinephrine infusion intermittantly pre and post intervention
- Acetaminophen Group: TOTAL: 5 stable febrile (temp >38.3°C) ICU patients/participants.
  Acetaminophen: one-time dose of acetaminophen 650mg given via the enteral route (via the gut) after which vital signs (including continuous measures of core temperature, heart rate, and blood pressure) will be monitored for 4 hours.
  Only 1 of the 5 participants were receiving any vasoactive infusions. The one participant was receiving low dose milrinone that was weaned off in the post intervention period. There was no conversion to equivalent dose of norepinephrine.
Arm/Group | Control Group | Acetaminophen Group
Number analyzed (Participants) | 1 | 1
mcg
  Pre-Intervention (2 hours) TOTAL Norepinephrine | 167.0 | NA — None given during this period
  Pre-Intervention (2 hours) TOTAL Milrinone | NA — None given during this period | 6000.0
  Post-Intervention (4 hours) TOTAL Norepinephrine | 576.0 | NA — None given during this period
  Post-Intervention (4 hours) TOTAL Milrinone | NA — None given during this period | 7000.0

4. Secondary Outcome: Equivalent-volume Fluid Administered Post Intervention
Description: Total crystalloid and colloid fluid will be converted the the equi-volume dose (with the ratio 1.4:1 (as per Finfer et al.(2004) & Vincent and Weil (2006) before making comparisons between the treatment and control groups.
Time Frame: 4 hours post intervention
Measure: Mean (Full Range); unit: mL
Arm/Group | Control Group | Acetaminophen Group
Number analyzed (Participants) | 1 | 5
mL
  Pre-Intervention (2 hours) Total fluid INTAKE | 235 [235 to 235] | 298 [30 to 736]
  Pre-Intervention (2 hours) Total fluid OUTPUT | 80 [80 to 80] | 370 [140 to 790]
  Post-Intervention (4 hours) Total Fluid INTAKE | 734 [734 to 734] | 612 [353 to 856]
  Post-Intervention (4 hours) Total Fluid OUTPUT | 245 [245 to 245] | 852 [230 to 1400]

5. Secondary Outcome: Fever Burden
Description: Continuous measurements of core body temperature will be recorded for 6 hours. Fever burden (FB) is defined as area between the 6 hour temperature curve and 38.3°C cut-off and it is reported in °C-hour.
  PRE-INTERVENTION FB: is reported for a 2 hour period. POST-INTERVENTION FB: post-intervention fever burden is reported for a 6 hour period and average hourly fever burden.
  Peak Temperature: is the highest recorded temperature for the study period in °C Minimum Temperature: is the lowest recorded temperature for the study period in °C
Time Frame: 6 hours post intervention
Population: NOTE: there was some data loss for the one participant in the control group. Temperature was recorded every 5 minutes for the first 40 minutes and then only hourly due to technical failure which may impact the accuracy of fever burden calculations.
Measure: Mean (Full Range); unit: °C*hours
Arm/Group | Control Group | Acetaminophen Group
Number analyzed (Participants) | 1 | 5
°C*hours
  Pre-Intervention FB (2 hours) | 0.97 [0.97 to 0.97] | 2.16 [1.07 to 3.78]
  Post-Intervention FB (6 hours) | 0.74 [0.74 to 0.74] | 5.65 [1.60 to 10.24]

ADVERSE EVENTS:
Time Frame: Until ICU discharge (max 28 days)
Arm/Group | Control Group | Acetaminophen Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/5
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/5
Other Adverse Events (participants affected / at risk) | 0/1 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No